CLINICAL TRIAL: NCT05179837
Title: Early Feasibility Study of Endoscopic Optical Coherence Tomography for Screening and Diagnosis of Colorectal Precancerous and Malignant Polyps
Brief Title: Endoscopic Optical Coherence Tomography for Screening and Diagnosis of Colorectal Precancerous and Malignant Polyps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202103151
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer; Rectal Cancer; Cancer of the Rectum; Cancer of the Colon; Precancerous Polyp; Malignant Polyp
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Optical coherence tomography (OCT) probe (Experimental): After consent, the endoscopist will perform a standard of care colonoscopy. If a polyp is found, then OCT will be used to image that polyp. Patients with polyps, regardless of number found, will have either one tubular adenoma (NICE type 2) imaged OR one hyperplastic polyp (NICE type 1) imaged. If no polyps are found, then one area of normal mucosa will be imaged. If on the rare chance a malignant appearing colonic tumor (NICE type 3) is found, this and no other polyps will be imaged with OCT.
  Interventions: Device: Optical coherence tomography probe

INTERVENTIONS:
Device: Optical coherence tomography probe — The OCT probe is attached to an approximately 3-meter wire that is attached to the OCT fiber probe system setup. This setup consists of a power supply unit, and a control platform that controls fiber probe rotation and retraction. The OCT probe will be advanced through the colonoscope instrument channel
  Other Names: OCT probe

SUMMARY:
Colorectal cancer arises from the mucosal layer of the colon. Current screening is performed by flexible endoscopy, which involves visual inspection of the mucosal lining of the colon and rectum with an optical camera mounted on the endoscope, with abnormal areas being biopsied. This method is somewhat limited in that there are no readily available surface pattern or morphological classification systems with adequate sensitivity or specificity to evaluate extent of submucosal invasion (deep, superficial, or none). Optical coherence tomography (OCT) using pattern recognition is a high-resolution imaging modality. There is currently an unmet need to predict depth of invasion for colonic tumors to decide on applicability of endoscopic (endoscopic submucosal dissection or endoscopic mucosal resection) vs. surgical therapy. The investigators' hypothesis is that OCT will have a higher diagnostic accuracy for determining depth of submucosal invasion compared to existing modalities. The investigators will first aim to assess the procedural feasibility and safety of using an OCT probe during routine colonoscopy with an early feasibility study. This study will identify appropriate modifications to the device and help with development of subsequent clinical study protocols. The eventual goal is to assess the diagnostic accuracy of OCT imaging for predicting depth of invasion of colonic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing standard of care colonoscopy for the evaluation of colonic polyps.
* At least 40 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Pregnant and/or breastfeeding.
* Unable to tolerate sedation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kushnir, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optical Coherence Tomography (OCT) Probe
Started | 36
Completed | 32
Not Completed | 4
Not completed — Lesion turned out to be scar tissue and not a polyp | 1
Not completed — Device malfunctioned | 1
Not completed — Image quality too low | 2

BASELINE CHARACTERISTICS:
Arm/Group | Optical Coherence Tomography (OCT) Probe
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 64.5 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Whose Procedure Length Using an OCT Probe During Routine Colonoscopy is Within 5 Minutes
Description: If the proportion of the patients whose procedure length using an OCT probe during routine colonoscopy is within 5 minutes is greater than 75%, then the feasibility is defined in this study.
Time Frame: Within 5 minutes during standard of care colonoscopy - Day 1 (average length 3:40 minutes (full range 1:54-8:20 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Optical Coherence Tomography (OCT) Probe
Number analyzed (Participants) | 35
Participants | 29

2. Secondary Outcome: Number of Participants With Adverse Events Related to OCT Imaging During Routine Colonoscopy
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: From start of colonoscopy through 48 hours after colonoscopy (estimated time of 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Optical Coherence Tomography (OCT) Probe
Number analyzed (Participants) | 35
Participants | 0

3. Secondary Outcome: Number of Participants Who Have a Successfully Captured OCT Image Using Machine Learning Algorithm
Description: Whether OCT image is successfully captured using machine learning algorithm, coded as "good" or "noisy".
Time Frame: During colonoscopy (Day 1)
Population: 4 participants were excluded due to absence of polyps (n=1), probe malfunction (n=1), and poor image quality (n=2).
Measure: Count of Participants; unit: Participants
Arm/Group | Optical Coherence Tomography (OCT) Probe
Number analyzed (Participants) | 32
Participants | 32

4. Secondary Outcome: Cohen's Weighted Kappa Score
Description: Overall agreement (OCT probe yielding results consistent with clinical pathology biopsy results) as measured by Cohen's Kappa. Overall Cohen's Kappa is a statistical measure for assessing the reliability of agreement between the two results by taking into account the element of chance. Cohen's kappa can range from 0 to 1 with 1 indicating perfect agreement and 0 indicating an agreement equivalent to chance.
  Clinical pathology is the gold standard for diagnosis. Diagnosis from both OCT and clinical pathology will be assigned as normal mucosa, hyperplastic polyp, tubular adenoma, sessile serrated adenoma, or colorectal cancer.
Time Frame: During colonoscopy (Day 1)
Population: 4 participants were excluded due to absence of polyps (n=1), probe malfunction (n=1), and poor image quality (n=2).
Measure: Number (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Optical Coherence Tomography (OCT) Probe
Number analyzed (Participants) | 32
proportion of agreement | 0.845 [0.774 to 0.915]

ADVERSE EVENTS:
Time Frame: From start of colonoscopy through 48 hours after colonoscopy (estimated time of 3 days).
Arm/Group | Optical Coherence Tomography (OCT) Probe
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optical Coherence Tomography (OCT) Probe (N=35)
Palpitations (Cardiac disorders) | 1
Potential statin myopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 2
Ileal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Right arm pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhagic shock (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT05179837/Prot_SAP_000.pdf